CLINICAL TRIAL: NCT03346668
Title: Role of Neurogenic Inflammation and Topical 6% Gabapentin Therapy in Symptomatic Scarring Alopecia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110336
Record Dates: First submitted 2017-09-08; First posted 2017-11-17 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Scarring Alopecia; Frontal Fibrosing Alopecia; Lichen Planopilaris; Central Centrifugal Cicatricial Alopecia; Central Centrifugal Scarring Alopecia
MeSH Terms: conditions — Alopecia; Lichen Planus | interventions — Gabapentin; Solutions

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Topical gabapentin (Experimental): gabapentin 6% solution, 1mL applied twice daily for 12 weeks
  Interventions: Drug: Topical gabapentin

INTERVENTIONS:
Drug: Topical gabapentin — topical gabapentin 6% solution
  Other Names: gabapentin 6% solution

SUMMARY:
This study will serve as a pilot study to determine the efficacy and safety of topical gabapentin in the treatment of symptomatic scarring alopecia.

DETAILED DESCRIPTION:
Primary scarring alopecias (PSAs) are poorly understood dermatologic disorders that result in permanent hair loss. Most of the scarring alopecias involve a painful course, with individuals reporting scalp pain, burning, itching, or tingling/crawling sensations that can ultimately impact physical and psychological health. There has been no study of topical neurogenic agents, such as gabapentin, to treat scarring alopecia. However topical gabapentin has been safely used in other conditions associated with chronic pain, burning, irritation, itch, or tingling, such as vulvodynia. This study will serve as a pilot study to determine the efficacy and safety of topical gabapentin in the treatment of symptomatic scarring alopecia. In this study, 10 subjects with symptomatic lymphocytic-type scarring alopecia will be recruited and treated with topical gabapentin. Disease burden will be evaluated before and after 12 weeks of treatment through reporting of subjective symptomatology via surveys/questionnaire, neurometer study, clinical assessment, and biopsies measuring levels of CGRP before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults, greater than 18 years of age
2. Biopsy-proven diagnosis of primary scarring alopecia of lymphocytic inflammatory infiltrate type, indicated as one of the following conditions: lichen planopilaris, frontal fibrosing alopecia, or central centrifugal cicatricial alopecia
3. At least one persistent scalp symptom associated with inflammation: pain, burning, itch, tingling/crawling, stinging, or tenderness
4. Able to complete survey and questionnaire subjectively
5. Consents to participate in neurometer study and scalp biopsy acquisition
6. Willingness to adhere to study protocol
7. If subject is taking a neuromodulatory medication (including capsaicin cream, tricyclic antidepressants, carbamazepine, phenytoin, topiramate, oxcarbazepine, lamotrigine, morphine, Botox, etc), he or she must be a stable dose for at least 6 months prior to study enrollment

Exclusion Criteria:

1. Allergy or intolerance to gabapentin or the substances used in its compounding
2. Underlying disease that might be adversely affected by topical gabapentin
3. Application of topical immunomodulatory or immunosuppressive agent to the scalp in the preceding 2 weeks
4. Systemic administration of corticosteroid or other systemic treatment (i.e., methotrexate, phototherapy) that has immunomodulatory or other immunosuppressive mechanism of action, in the preceding 8 weeks
5. Clinical evidence of secondary skin infection
6. Individuals who have undergone scalp reduction surgery or hair transplantation
7. Asymptomatic disease
8. Immunosuppression due to disease state or use of systemic/topical biological agents (HIV, chemotherapy, immunomodulators, history of transplantation)
9. Any Investigational medications within the past 30 days, including those for migraines or scarring alopecias (anti-CGRP agents)
10. Use of GABAergic medications (including gabapentin and pregabalin) in the preceding 2 months
11. Use of illicit drugs or opioid medications
12. Evidence of anemia, thyroid disease, sarcoidosis or other medical condition that could impact hair growth and adversely impact the outcome of the study
13. Implantable Cardioverter Defibrillator (ICD) or pacemaker
14. Subject has any medical condition that, in the judgment of the Investigator, would jeopardize the subject's safety following exposure to the administered medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Neurogenic inflammation-QOL | Change from Baseline to 14 weeks
  Complete a QOL (Quality of Life) survey Scale= (Not relevant to Extremely Relevant)
Neurogenic inflammation-Short Form (36) Health Survey | Change from Baseline to 14 weeks
  Complete Short Form (36) Health Survey Scale Scale=1-5 1 being the best and 5 being the worse
Neurogenic inflammation- Visual Analog pain Scale | Change from Baseline to 14 weeks
  Visual Analog Pain scale Scale = 1-10 1 being the least pain and 10 being the worse pain

SECONDARY OUTCOMES:
Safety and efficacy of topical 6% gabapentin -Medication side Effects | Change from Baseline to 12 weeks
  Subjects will have Medication side effects collected at day 0 and ending week 12
Safety and efficacy of topical 6% gabapentin -Blood levels | Change from Baseline to 12 weeks
  Subjects will have blood levels measured at Day 0 and 12 weeks
Safety and efficacy of topical 6% gabapentin -Adverse Events | Change from Baseline to 12 weeks
  Subjects will have adverse events collected on day 0 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-01-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT03346668/Prot_000.pdf